CLINICAL TRIAL: NCT00823810
Title: Treatment Monitoring of Advanced Colorectal Cancer With 18F-FDG PET/CT
Acronym: RESCORE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment promlems
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Marko Seppanen, MD, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RESCORE
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Response to treatment; FDG PET/CT
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Colorectal cancer (Experimental)
  Interventions: Other: PET/CT

INTERVENTIONS:
Other: PET/CT — 18F-FDG PET/CT

SUMMARY:
Measuring tumor response to treatment based on computed tomography (CT) and/or magnetic resonance imaging (MRI) has been a widely debated issue (response criteria in solid tumors [RECIST] and World Health Organization criteria). Furthermore, early identification of nonresponding patients is of great importance because the rates of response of common malignant solid tumors to chemotherapy are in the range of only 20-30%. Therefore, quantitative imaging of tumor metabolism with 18F-FDG PET/CT may provide important advantages and thus reduce side effects and costs of ineffective therapy. However, the evidence to date for the use of 18F-FDG-PET/CT with this indication is limited.

The purpose of the present trial is to determine the impact of 18F-FDG PET/CT in the management of advanced colorectal cancer. The aim is also to confirm whether a metabolic response can be used as a surrogate end point in monitoring treatment response in this cancer type.

The study consists of 40 patients with advanced colorectal cancer patients. All patients will be studied with 18F-FDG PET/CT combined with diagnostic contrast enhanced abdominal CT before the start of chemotherapy and re-evaluated 4-5 weeks after the initiation of therapy. Effect of this metabolic and anatomic change in therapy are evaluated and correlated to survival, morbidity, and treatment -related costs. Histopathologic confirmation of response is evaluated whenever possible. The data will be collected between 2008 and 2012.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 80 years old
* Language spoken: Finnish or Swedish
* Performance status: Karnofsky score 70 or better or WHO performance status 2 or better
* earlier diagnosed (histologically confirmed) colorectal cancer with discovered metastases at operation
* Earlier diagnosed and treated colorectal cancer with discovered recurrence in the follow up
* Mental status: Patients must be able to understand the meaning of the study
* Informed consent: The patient must sign the appropriate Ethical Committee (EC) approved informed consent documents in the presence of the designated staff

Exclusion Criteria:

* Prior medical history: Patient must have no history of serious cardiovascular, liver or kidney disease
* Vulnerable study subjects such as described in Finnish law concerning clinical studies (disabled, children, pregnant or breast-feeding women, prisoners) will not be included.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Survival | 2 years

SECONDARY OUTCOMES:
Time to progression | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland

REFERENCES:
- See also: Turku PET Centre — http://www.turkupetcentre.fi/